CLINICAL TRIAL: NCT06317597
Title: Evaluating the Efficacy of Short Time Intervals in Split-Dose Bowel Preparation of Oral Sulfate Solution: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Efficacy of Short Time Intervals in Split-Dose Bowel Preparation of Oral Sulfate Solution for Colonoscopy
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Suzhou Hospital of Nanjing Medical University (Unknown); Tianjin First Central Hospital (Other); Tianjin Beichen Hospital (Unknown); Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); First People's Hospital of Hangzhou (Other); The Third People's Hospital of Chengdu (Other); Ningbo Yinzhou District Second Hospital (Unknown); Changshu Affiliated Hospital of Soochow University (Other); Linyi People's Hospital (Other); Shanghai East Hospital (Other); Heilongjiang Province Hospital Nangang Branch (Unknown); The Affiliated Jiangyin Hospital of Nantong University (Unknown); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OSS2024-0311
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Colonoscopy: Bowel Preparation
Keywords: time interval; bowel preparation; Oral Sulfate Solution（OSS）

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short time interval group: (Experimental): Bowel preparation for colonoscopy was performed using oral sulfate solution as a laxative
  Interventions: Drug: Magnesium Sulfate，Sodium Sulfate and Potassium Sulfate Concentrate Oral Solution
- Standard time interval group (Active Comparator): Bowel preparation for colonoscopy was performed using oral sulfate solution as a laxative
  Interventions: Drug: Magnesium Sulfate，Sodium Sulfate and Potassium Sulfate Concentrate Oral Solution

INTERVENTIONS:
Drug: Magnesium Sulfate，Sodium Sulfate and Potassium Sulfate Concentrate Oral Solution — OSS contained 17.5 g sodium sulfate, 3.13 g potassium sulfate, 1.6 g magnesium sulfate, and flavoring agents in an aqueous liquid form supplied in a 177 mL bottle. Dilute 177ml sodium, potassium, and magnesium sulfate oral solution to 500ml and intake 12-14 hours before colonoscopy, followed by two doses of 500ml water or clear aqueous liquid within 2 hours; Repeat the procedure 6 hours before the colonoscopy.
  Arms: Short time interval group:
Drug: Magnesium Sulfate，Sodium Sulfate and Potassium Sulfate Concentrate Oral Solution — OSS contained 17.5 g sodium sulfate, 3.13 g potassium sulfate, 1.6 g magnesium sulfate, and flavoring agents in an aqueous liquid form supplied in a 177 mL bottle. Dilute 177ml sodium, potassium, and magnesium sulfates oral solution to 500ml and intake 16-18 hours before the colonoscopy, followed by two doses of 500ml water or clear aqueous liquid within 2 hours; Repeat the procedure 6 hours before the colonoscopy.
  Arms: Standard time interval group

SUMMARY:
To evaluate whether oral sulfate solution administered in a short time interval (6-8 hours) between the first and last dose of laxative is not inferior to a long time interval (10-12 hours) in bowel preparation quality.

DETAILED DESCRIPTION:
The split-dose bowel preparation is recommended by multiple guidelines and widely used worldwide for improved bowel preparation quality, higher detection rate of colorectal lesions, and better tolerance. The effect of the time interval between the last dose of laxative and the colonoscopy on the quality of bowel preparation has been well studied, but the impact of the time interval between the first and last dose of laxative on the bowel preparation quality deserve to be explored. Oral sulfate solution administered in a short time interval can reduce sleep disturbance and hunger and is more flexible and convenient. This study aims to evaluate whether oral sulfate solution administered in a short time interval (6-8 hours) is not inferior to a long time interval (10-12 hours) on bowel preparation quality.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign informed consent;
* Subjects who require screening, surveillance, and diagnostic colonoscopy;
* Subjects who take the oral sulfate solution for bowel preparation.

Exclusion Criteria:

* Subjects with serious cardiac and cerebrovascular diseases, bronchial and lung diseases, suffering from metabolic disease or endocrine disease, abnormal blood clotting mechanism, malignant tumor, electrolyte abnormalities, epilepsy, renal or liver dysfunction;
* Subjects with ascites, suspected electrolyte abnormalities, or uncorrected dehydration.
* Subjects with confirmed or suspected gastrointestinal obstruction, gastric retention, gastroparesis, gastric emptying disorder, or acute gastrointestinal bleeding;
* Subjects with confirmed or suspected colorectal cancer, inflammatory bowel disease, toxic colitis, or toxic megacolon.
* Subjects who had previously undergone colorectal resection.
* Subjects with constipation or suspected severe gastric motility disorder;
* Women with positive pregnancy tests or pregnancy plans, and women in lactation;
* Subjects who have participated in any other clinical trials within the last 3 months;
* Subjects with any other conditions that the investigator considered inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation adequate rate | 30minutes
  Adequate bowel cleansing was defined as a total Boston Bowel Preparation Scale (BBPS) ≥ 6 with a partial BBPS ≥ 2 in each colon segment.

SECONDARY OUTCOMES:
Acceptability of bowel preparation by questionnaire survey | 12 hours

OTHER OUTCOMES:
Incidence of laxative-related adverse events assessed by clinical examinations | 8 days
Colonoscopy completion rate | 30 minutes
  Proportion of subjects receiving complete colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No